CLINICAL TRIAL: NCT00397501
Title: A Phase I/II Pilot Study of Patients With Brain Metastasis Secondary to Breast Cancer Treated With Methotrexate and Carboplatin in Conjunction With Blood-Brain Barrier Disruption, With Concurrent Trastuzumab in HER-2 Positive Patients
Brief Title: BBBD Followed By Methotrexate and Carboplatin With or Without Trastuzumab in Treating Women With Breast Cancer That Has Spread to the Brain
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: after original approval, IRB closed enrollment; major revisions required to re-open.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002188; 2188 (Other: OHSU eIRB); SOL-06015 (Other: OHSU Knight Cancer Institute); OHSU-2188 (Other: OHSU IRB)
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Brain and Central Nervous System Tumors; Breast Cancer; Cognitive/Functional Effects; Drug/Agent Toxicity by Tissue/Organ; Psychosocial Effects of Cancer and Its Treatment
Keywords: cognitive/functional effects; psychosocial effects of cancer and its treatment; drug/agent toxicity by tissue/organ; recurrent breast cancer; stage IV breast cancer; adult tumors metastatic to brain
MeSH Terms: conditions — Central Nervous System Neoplasms; Breast Neoplasms; Drug-Related Side Effects and Adverse Reactions; Brain Neoplasms | interventions — Trastuzumab; Carboplatin; Methotrexate; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HER-2 positive subjects (Active Comparator): HER-2 positive subjects treated with trastuzumab
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: methotrexate; Drug: sodium thiosulfate
- HER-2 negative subjects (Active Comparator): HER-2 negative subjects not treated with trastuzumab
  Interventions: Drug: carboplatin; Drug: methotrexate; Drug: sodium thiosulfate

INTERVENTIONS:
Biological: trastuzumab — Trastuzamab, 6mg/kg, within 48 hrs before BBBD
  Then, Trastuzumab, 2mg/kg, weekly until next BBBD Then continue for 12 cycles
  Other Names: Herceptin
  Arms: HER-2 positive subjects
Drug: carboplatin — 200mg/m2/day x 2 days; total dose 400mg/m2 Infused i.a. over 10 mins in 200ml of normal saline after MTX infusion
  Other Names: carbo
Drug: methotrexate — 2500 mg/day x 2 days; total dose 5000mg Infused over 10mins in 200ml saline beginning immediately after mannitol infusion
  Other Names: MTX
Drug: sodium thiosulfate — STS dose admin i.v. over 15mins @ 4hrs post carboplatin = 20gm/m2; STS dose admin i.v. over 15mins @ 8hrs post carboplatin = 16gm/m2
  Other Names: STS

SUMMARY:
RATIONALE: Osmotic blood-brain barrier disruption uses certain drugs, such as mannitol, to open the blood vessels around the brain and allow tumor-killing substances to be carried directly to the brain. Drugs used in chemotherapy, such as methotrexate and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Trastuzumab may also help methotrexate and carboplatin work better by making tumor cells more sensitive to the drugs. Giving osmotic blood-brain barrier disruption together with methotrexate, carboplatin, and trastuzumab may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of carboplatin when given together with methotrexate and trastuzumab after mannitol in treating women with breast cancer that has spread to the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and toxicity associated with blood-brain barrier disruption comprising transfemoral mannitol followed by methotrexate and carboplatin with or without trastuzumab (Herceptin®) in women with brain metastasis secondary to breast cancer. (Phase I)
* Determine if overall survival exceeds 5 months in patients with Human Epidermal growth factor Receptor 2(HER2)-positive or HER2-negative disease treated with this regimen. (Phase II)

Secondary

* Determine the overall survival of these patients.
* Compare the event-free and overall survival, steroid use, response rates, and time to best response in patients with HER2-positive vs HER2-negative disease.
* Assess the quality of life of patients treated with this regimen.
* Assess the neuropsychological effects of this treatment regimen in these patients.
* Determine cerebrospinal fluid levels of trastuzumab before and after blood-brain barrier disruption.

OUTLINE: This is a multicenter, phase I, pilot, dose-finding study of carboplatin followed by a phase II, open-label study.

* Phase I: Patients undergo osmotic blood-brain barrier disruption (BBBD) comprising mannitol by transfemoral catheterization followed by methotrexate intra-arterially (IA) over 10 minutes and carboplatin IA over 10 minutes on days 1 and 2. Patients also receive sodium thiosulfate IV over 15 minutes at 4 and 8 hours after each dose of carboplatin; leucovorin calcium IV or orally every 6 hours on days 3-9; and pegfilgrastim subcutaneously (SC) on day 4 or filgrastim (G-CSF) SC beginning on day 4 and continuing until blood counts recover (7-10 days). Patients with HER-2 positive disease receive trastuzumab (Herceptin®) IV over 90 minutes within 48 hours prior to BBBD and then weekly for 3 weeks (between BBBD therapy sessions). Treatment repeats every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive decreasing doses of carboplatin and/or methotrexate if the proposed dose is not well tolerated. Dose-limiting toxicity is defined as grade IV hematologic toxicity with delay in subsequent treatment courses for 4 weeks OR grade III/IV nonhematologic toxicity without recovery in 14 days during the course of treatment.

* Phase II: Patients undergo BBBD as in phase I and receive carboplatin and methotrexate at the doses determined in phase I. Patients also receive sodium thiosulfate, leucovorin calcium, and pegfilgrastim or G-CSF as in phase I. Patients with HER2-positive disease also receive trastuzumab as in phase I.

Neuropsychological assessment is performed at baseline, every 6 months during treatment, every 6 months for 1 year, and then annually thereafter. Quality of life is assessed at baseline, every 3 months during treatment, at the completion of study treatment, every 6 months for 1 year, and then annually thereafter.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 78 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer metastatic to the central nervous system (as documented by brain biopsy, cytology [analysis from cerebrospinal fluid]) OR radiographic evidence of brain metastasis with a diagnosis of systemic breast cancer
* Patients must have stable or no systemic disease as determined by a CT scan of the chest, abdomen, and pelvis
* HER2-positive or -negative disease by fluorescent in situ hybridization (FISH) or immunohistochemistry
* Patients with HER2-positive disease and signs of intracranial herniation and/or spinal block may first undergo intraarterial chemotherapy off study (with carboplatin, methotrexate, and trastuzumab [Herceptin®] by the same routes used on study) until radiographically shown to be safe to undergo blood brain barrier disruption, at which point they may be enrolled in the study
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 6 weeks
* Hematocrit ≥ 25%
* WBC ≥ 2,500/mm³
* Absolute neutrophil count ≥ 1,200/mm³
* Platelet count ≥100,000/mm³
* Creatinine clearance ≥ 50 mL/min (eligible for full-dose methotrexate) (30-49 mL/min allowed for patients receiving reduced-dose methotrexate)
* Bilirubin ≤ 2.0 times upper limit of normal
* LVEF normal by echocardiogram or MUGA
* Adequate pulmonary and cardiac function to tolerate general anesthesia as determined by physical examination and history
* No New York Heart Association class III-IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known allergy to trastuzumab (HER2-positive patients), carboplatin, methotrexate, or sodium thiosulfate
* No hepatitis B or C positivity
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection (e.g., HIV)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* Prior surgery or biopsy allowed
* Prior chemotherapy and radiation therapy for metastatic breast cancer allowed
* No radiation or cytotoxic chemotherapy within the past 4 weeks (except trastuzumab or hormone therapy that has been part of the patient's ongoing treatment [e.g., aromatase inhibitors for estrogen receptor positive patients])
* No noncytotoxic regimens (e.g., targeted oral agents) within the past 2 weeks
* No investigational agents within the past 4 weeks
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival exceeding 5 months in patients with Human Epidermal growth factor Receptor 2(HER2)-negative disease | 1 year after initiation of treatment
Overall survival exceeding 5 months in patients with HER2-positive disease | 1 year after initiation of treatment

SECONDARY OUTCOMES:
Overall survival | 5 years after intitiation of treatment
Progression-free survival | 5 years
Complete response rate | 5 years
Time to best response | 5 years
Quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Neuwelt, MD, Principal Investigator — OHSU Knight Cancer Institute